CLINICAL TRIAL: NCT04442789
Title: Long-term Sequelae of Severe Sars-CoV-2 Infections
Brief Title: Sequelae of Sars-CoV-2 Infections
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: SECOV
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Lung Diseases; Cardiac Disease; Inflammatory Reaction
MeSH Terms: conditions — Lung Diseases; Heart Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMCs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By the end of 2019 a new coronavirus, named SARS-CoV-2, was discovered in patients with pneumonia in Wuhan, China. In the following weeks and months the virus spread globally, having a tremendous impact on global health and economy. To date, no vaccine or therapy is available. Severe courses of the infection not only affect the lungs, but also other organs like the heart, kidney, or liver. The lack of preexisting immunity might at least partially explain the affection of extra pulmonary organs not yet seen in infections due to other respiratory viruses. In this observational investigation the study group will follow up on patients that have been hospitalized due to a SARS-CoV-2 infection, and monitor sequelae in various organs, with an emphasis on the pulmo-cardiovascular system. Our that in some patients, organ damage will persist and require long-term medical care.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) caused by SARS-CoV-2 requires hospitalization in a significant amount of patients. The hospitalization rate and disease severity increases in the elderly and patients with comorbidities such as diabetes, arterial hypertension, lung pathologies and obesity (Garg et al.). Patients with severe infections have pneumonia, requiring prolonged invasive ventilation. Sequelae of longer periods of mechanical ventilation and reduction of quality of life after acute respiratory distress syndrome (ARDS) are described (Herridge et al., 2 references). Besides, SARS-CoV-2 can induce - without preexisting immunity - strong inflammatory reactions, which can affect various organs. COVID-19 specific complications like thromboembolic events, neurologic events, myocardial involvement, or liver damage are reported during the acute stage of the infection. The lung is affected even during less severe infections, and ground glass opacities can result in consolidations (Shi et al.). These changes were reported to persist after discharge (Mo et al.). Acute kidney failure occurs in critically ill patients in 20-40% (Richardson et al.), and 40% of patients admitted to the hospital had proteinuria (Cheng et al.). Myocardial damage is reported, and some patients even presented initially with chest tightness and palpitations before having fever or cough (Zheng et al.). Moreover, patients with COVID-19 have a higher risk of thromboembolic events (Klok et al., Llitjos et al). Typically these patients have a prolonged activated partial thromboplastin time (aPTT), and often antiphospholipid antibodies (Bowles et al.). The long-term consequences of the strong inflammatory response affecting various organs are currently unknown. We hypothesize that some patients will have transient or persistent sequelae requiring medical care. The study group will therefore clinically examine patients that were hospitalized due to COVID-19, and monitor pulmonary, and other organ functions for at least one year after symptom onset. The study group will thereby perform lung and cardial examinations, monitor nephrologic parameters and perform radiology. Pneumologic tests will include a lung function test, a spiroergometry, a 6-minute walking test, and a grip-force test. Cardiac examination will include an echocardiography, and an electrocardiogram. In case of of severe pneumonia, or deterioration in lung function, computer tomography of the lungs will be performed. Blood (and urine) tests will include kidney parameters, inflammatory markers, liver values, and coagulation tests. Additional examinations will be done on an individual basis if clinically indicated, e.g. lung biopsies in case of suspected interstitial fibrosis. Additionally patient samples, which were taken for diagnostic purposes (serum, PBMCs, biopsies) will be stored in the biobank of the German center for lung research (DZL). Clinical evaluation and testing will start 2 months after symptom onset and the last visit is scheduled 10 months later. Depending on the results and the needs of the individual patient additional testing will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* hospitalization due to Sars-CoV-2 infection

Exclusion Criteria:

* under 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients that have been hospitalized due to Covid 19
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sequelae after COVID-19 | 12 months, extension if required
  Identify organ dysfunction after SARS-CoV-2 infections

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine II, Universities of Giessen and Marburg Lung Center (UGMLC), member of the German Center for Lung Research (DZL), Justus-Liebig-University, Giessen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garg S, Kim L, Whitaker M, O'Halloran A, Cummings C, Holstein R, Prill M, Chai SJ, Kirley PD, Alden NB, Kawasaki B, Yousey-Hindes K, Niccolai L, Anderson EJ, Openo KP, Weigel A, Monroe ML, Ryan P, Henderson J, Kim S, Como-Sabetti K, Lynfield R, Sosin D, Torres S, Muse A, Bennett NM, Billing L, Sutton M, West N, Schaffner W, Talbot HK, Aquino C, George A, Budd A, Brammer L, Langley G, Hall AJ, Fry A. Hospitalization Rates and Characteristics of Patients Hospitalized with Laboratory-Confirmed Coronavirus Disease 2019 - COVID-NET, 14 States, March 1-30, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 17;69(15):458-464. doi: 10.15585/mmwr.mm6915e3. PMID 32298251
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Shi H, Han X, Jiang N, Cao Y, Alwalid O, Gu J, Fan Y, Zheng C. Radiological findings from 81 patients with COVID-19 pneumonia in Wuhan, China: a descriptive study. Lancet Infect Dis. 2020 Apr;20(4):425-434. doi: 10.1016/S1473-3099(20)30086-4. Epub 2020 Feb 24. PMID 32105637
- [Background] Mo P, Xing Y, Xiao Y, Deng L, Zhao Q, Wang H, Xiong Y, Cheng Z, Gao S, Liang K, Luo M, Chen T, Song S, Ma Z, Chen X, Zheng R, Cao Q, Wang F, Zhang Y. Clinical Characteristics of Refractory Coronavirus Disease 2019 in Wuhan, China. Clin Infect Dis. 2021 Dec 6;73(11):e4208-e4213. doi: 10.1093/cid/ciaa270. PMID 32173725
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Cheng Y, Luo R, Wang K, Zhang M, Wang Z, Dong L, Li J, Yao Y, Ge S, Xu G. Kidney disease is associated with in-hospital death of patients with COVID-19. Kidney Int. 2020 May;97(5):829-838. doi: 10.1016/j.kint.2020.03.005. Epub 2020 Mar 20. PMID 32247631
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Background] Bowles L, Platton S, Yartey N, Dave M, Lee K, Hart DP, MacDonald V, Green L, Sivapalaratnam S, Pasi KJ, MacCallum P. Lupus Anticoagulant and Abnormal Coagulation Tests in Patients with Covid-19. N Engl J Med. 2020 Jul 16;383(3):288-290. doi: 10.1056/NEJMc2013656. Epub 2020 May 5. No abstract available. PMID 32369280
- [Derived] Kimmig LM, Rako ZA, Ziegler S, Richter MJ, G S AT, Roller F, Grimminger F, Vadasz I, Seeger W, Herold S, Tello K, Matt U. Long-term comprehensive cardiopulmonary phenotyping of COVID-19. Respir Res. 2022 Sep 21;23(1):263. doi: 10.1186/s12931-022-02173-9. PMID 36131349